CLINICAL TRIAL: NCT03599713
Title: A Phase 2 Study of INCMGA00012 in Participants With Metastatic Merkel Cell Carcinoma (POD1UM-201)
Brief Title: A Study of INCMGA00012 in Metastatic Merkel Cell Carcinoma (POD1UM-201)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCMGA 0012-201; 2018-001627-39 (EudraCT Number)
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Merkel Cell Carcinoma
Keywords: Metastatic merkel cell carcinoma; anti-PD-1 antibody; immunoglobulin G4 (IgG4) monoclonal antibody; INCMGA00012
MeSH Terms: conditions — Carcinoma, Merkel Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Retifanlimab: Chemotherapy: Naïve (Experimental)
  Interventions: Drug: Retifanlimab
- Retifanlimab: Chemotherapy: Refractory (Experimental)
  Interventions: Drug: Retifanlimab

INTERVENTIONS:
Drug: Retifanlimab — INCMGA00012 administered at 500 milligrams (mg) by intravenous infusion once every 4 weeks
  Other Names: MGA012; INCMGA00012

SUMMARY:
The purpose of this study is to assess the clinical activity and safety of INCMGA00012 in participants with advanced/metastatic Merkel cell carcinoma (MCC).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Diagnosis of MCC with distant metastatic disease or recurrent, advanced locoregional disease not amenable to surgery or radiation
* Eastern Cooperative Oncology Group performance status of 0 to 1.
* Measurable disease according to RECIST v1.1.
* Availability of tumor tissue (fresh or archival) for central pathology review.
* Willingness to avoid pregnancy or fathering children based on protocol-defined criteria.

Exclusion Criteria:

* Prior systemic therapy for MCC, including chemotherapy and prior PD-1 or PD-L1-directed therapy.
* Treatment with anticancer drugs or participation in another interventional clinical study within 21 days before the first administration of study drug.
* Has not recovered to ≤ Grade 1 or baseline from toxic effects of prior therapy (with the exceptions for anemia not requiring transfusion support and any grade of alopecia) and/or complications from prior surgical intervention within 7 days before starting study treatment.
* Radiation therapy administered within 2 weeks of first dose of study treatment or radiation therapy to the thoracic region that is > 30 Gy within 6 months of the first dose of study treatment.
* Known central nervous system (CNS) metastases and/or carcinomatous meningitis.
* History of second malignancy within 3 years (with exceptions).
* Laboratory values outside the protocol-defined range at screening.
* Clinically significant pulmonary, cardiac, gastrointestinal or autoimmune disorders.
* Active bacterial, fungal, or viral infections, including hepatitis A, B, and C.
* Receipt of a live vaccine within 28 days of planned start of study therapy.
* Current use of protocol-defined prohibited medication.
* Known hypersensitivity to another monoclonal antibody that cannot be controlled with standard measures (eg, antihistamines and corticosteroids).
* Inability or unlikely, in the opinion of the investigator, to comply with the Protocol requirements.
* Participant who is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (65):
- United States (16):
  - Stanford Cancer Institute, Palo Alto, California
  - University of California San Francisco Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Rush University, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Mayo Clinic Rochester, Rochester, Minnesota
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of Nj, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Upmc Cancercenter, Pittsburgh, Pennsylvania
  - Inova Fairfax Hospital, Fairfax, Virginia
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia University Hospitals Inc, Morgantown, West Virginia
- St Vincent'S Hospital Sydney, Darlinghurst, New South Wales, Australia
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - Tom Baker Cancer Centre, Calgary AB, CA
  - London Health Sciences Centre Lhsc - South Street Hospital, London, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital Segal Cancer Ctr, Montreal, Quebec
  - McGill University Health Centre/Glen Site/Cedars Cancer Centre, Montreal, Quebec
- Czechia (4):
  - Fakultni Nemocnice Olomouc, Olomouc
  - Prof Mudr Petr Arenberger Drsc Mba, Prague
  - Nemocnice Na Bulovce, Prague
  - Thomayerova Nemocnice, Praha 4-krc
- France (7):
  - Hï¿½PITAL AMBROISE PAR, Boulogne-Billancourt
  - Chu Hopital de La Timone, Marseille
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hotel-Dieu, Nantes
  - CHU DE NICE - Hï¿½PITAL L'ARCHET 1, Nice
  - Hospital Saint Louis, Paris
  - HOPITAL CHARLES NICOLLE CHU ROUEN - Hï¿½PITAL DE BOIS-GUILLAUME, Rouen
  - Institut Gustave Roussy, Villejuif
- Germany (8):
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Elbe Klinikum Buxtehude, Buxtehude
  - Helios Klinikum Erfurt, Erfurt
  - Universitatsklinikum Essen, Essen
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Universitatsklinikum Giessen Und Marburg Gmbh, Klinik Für Innere Medizin, Marburg
  - University Hospital Regensburg, Regensburg
  - Universitaetsklinikum in Tubingen, Tübingen
- Hungary (3):
  - National Institute of Oncology, Budapest
  - Debreceni Egyetem Klinikai Kozpon Belgyogy Klinika, Debrecen
  - Szte Borgyogyszati Es Allergologiai Klinika, Szeged
- Italy (10):
  - Istituto Tumori Giovanni Paolo Ii Irccs Ospedale Oncologico Bari, Bari
  - Fondazione Del Piemonte Per L'Oncologia Ircc Candiolo, Candiolo
  - Irccs Azienda Ospedaliera Universitaria San Martino, Genova
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - European Institute of Oncology, Milan
  - A.O.U. Di Modena - Policlinico, Modena
  - Istituto Nazionale Tumori Irccs Fondazione Pascale, Naples
  - Iov - Istituto Oncologico Veneto Irccs, Padua
  - ONCOLOGIA ï¿½ IDI IRCCS ISTITUTO DERMOPATICO DELL'IMMACOLATA, Rome
  - Azienda Ospedaliera Universitaria Senese Policlinico Santa Maria Alle Scotte, Siena
- Centrum Onkologii - Instytut Im. Marii Sklodowskiej - Curie, Warsaw, Poland
- Spain (3):
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois (Chuv), Lausanne
  - Universitatsspital Zurich, Zurich
- United Kingdom (5):
  - Castle Hill Hospital, Cottingham
  - Royal Free London Nhs Foundation Trust, London
  - The Royal Marsden Nhs Foundation Trust, London
  - The Royal Marsden Nhs Foundation Trust - Sutton, Sutton
  - Royal Cornwall Hospital Truro Sunrise Centre, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grignani G, Rutkowski P, Lebbe C, Guida M, Gaudy-Marqueste C, Spagnolo F, Burgess M, Morano F, Montaudie H, Depenni R, Spada F, Yeung CCS, Pulini J, Cornfeld M, Tian C, Bhatia S. Phase II study of retifanlimab in patients with recurrent locally advanced or metastatic Merkel cell carcinoma (POD1UM-201). J Immunother Cancer. 2025 Aug 11;13(8):e012478. doi: 10.1136/jitc-2025-012478. PMID 40796223

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled and treated at 34 study centers in Italy, France, the United States, Poland, Canada, Switzerland, Hungary, the Czech Republic, Germany, Spain, and the United Kingdom.
Groups:
- Chemotherapy: Naïve: Participants with recurrent, advanced locoregional disease or distant metastatic disease who did not receive any prior chemotherapy received retifanlimab 500 milligrams (mg), administered by intravenous (IV) infusion over 60 minutes on Day 1 of each 28-day cycle (Q4W).
- Chemotherapy: Refractory: Participants with disease not responding to prior chemotherapy received retifanlimab 500 mg, administered by IV infusion over 60 minutes on Day 1 Q4W.
Period: Overall Study
Arm/Group | Chemotherapy: Naïve | Chemotherapy: Refractory
Started | 101 | 6
Safety Evaluable Population | 101 | 6
Enrolled Population | 101 | 6
Full Analysis Set | 65 | 6
Completed | 0 | 0
Not Completed | 101 | 6
Not completed — Death | 38 | 3
Not completed — Withdrawal by Subject | 17 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Discontinued Due to End of Study | 42 | 3

BASELINE CHARACTERISTICS:
Population: Baseline data were collected in members of the Safety Evaluable Population, comprised of all enrolled participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy: Naïve | Chemotherapy: Refractory | Total
Number analyzed (Participants) | 101 | 6 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (10.44) | 63.8 (10.46) | 70.7 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 1 | 34
  Male | 68 | 5 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 75 | 6 | 81
  Unknown or Not Reported | 25 | 0 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 78 | 6 | 84
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 22 | 0 | 22

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed overall response of complete response (CR) or partial response (PR), per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1), as determined by Independent Central Radiographic Review (ICR), at any post-Baseline visit until the first progressive disease (PD) or new anti-cancer therapy. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 26.8 months
Population: Full Analysis Set (FAS): all participants enrolled in the study who received at least 1 dose of study drug as of 15 October 2020 (selected to allow for at least 60 chemotherapy-naïve participants to be followed for at least 6 months after first response assessment). Analysis was based on the chemotherapy-naïve subset of the FAS. Confidence intervals (CIs) were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy: Naïve | Chemotherapy: Refractory
Number analyzed (Participants) | 65 | 0
percentage of participants | 52.3 [39.5 to 64.9] |

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from an initial objective response (CR or PR) per RECIST v1.1 until PD, or death due to any cause, as determined by ICR. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. A Kaplan-Meier estimate (estimated median) of the distribution function is reported.
Time Frame: up to 55.3 months
Population: Safety Evaluable Population: all enrolled participants who received at least 1 dose of study drug. Analysis was based on the chemotherapy-naïve subset of the population. Only those participants who had confirmed CR or PR prior to PD or start of new anticancer therapy were assessed. The 95% CI was calculated using the Brookmeyer and Crowley's method and Klein and Moeschberger's method with log-log transformation.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy: Naïve | Chemotherapy: Refractory
Number analyzed (Participants) | 55 | 0
months | NA [22.87 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. |

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a confirmed overall response (CR and PR) or stable disease (SD) (non-CR/non-PD) lasting at least 6 months from the start of treatment, until the first PD or new anti-cancer therapy, per RECIST v1.1 as determined by ICR. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions. PD: progression of a target or non-target lesion or presence of a new lesion. SD: no change in target lesions to qualify for CR, PR, or PD.
Time Frame: up to 57.1 months
Population: Safety Evaluable Population. Analysis was based on the chemotherapy-naïve subset of the population. CIs were calculated based on the exact method for binomial distributions.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy: Naïve | Chemotherapy: Refractory
Number analyzed (Participants) | 101 | 0
percentage of participants | 60.4 [50.2 to 70.0] |

4. Secondary Outcome: Progression-free Survival (PFS)
Description: According to RESIST v1.1, PFS was defined the time from the start of therapy until disease progression, or death due to any cause, as determined by ICR. Evaluation of target lesions: PD: ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. The sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered PD). Evaluation of non-target lesions: PD: Unequivocal progression of existing non-target lesions. (Note: the appearance of one or more new lesions is also considered PD).
Time Frame: up to 57.1 months
Population: Safety Evaluable Population. Analysis was based on the chemotherapy-naïve subset of the population. Median PFS time was estimated using the Kaplan-Meier method. The CI for median PFS time was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy: Naïve | Chemotherapy: Refractory
Number analyzed (Participants) | 101 | 0
months | 16.03 [9.03 to 32.23] |

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time in months between the first dose date (Day 1) and the date of death due to any cause.
Time Frame: up to 60.4 months
Population: Safety Evaluable Population. Analysis was based on the chemotherapy-naïve subset of the population. Median overall survival time was estimated using the Kaplan-Meier method. CI for median overall survival time was calculated using the method of Brookmeyer and Crowley.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy: Naïve | Chemotherapy: Refractory
Number analyzed (Participants) | 101 | 0
months | NA [45.24 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants died. |

6. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as either an AE reported for the first time or a worsening of a pre-existing event after the first dose of study drug until 90 days after the last dose of study drug. An AE with onset on/after starting a new anticancer therapy was not summarized as a TEAE.
Time Frame: up to 846 days (up to approximately 2.3 years)
Population: Safety Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy: Naïve | Chemotherapy: Refractory
Number analyzed (Participants) | 101 | 6
Participants | 92 | 5

7. Secondary Outcome: First-dose Cmax of Retifanlimab
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: preinfusion, 10 minutes postinfusion (± 10 minutes), and 4 hours postinfusion (± 10 minutes) on Day 1 of Cycle 1
Population: Pharmacokinetic (PK) Evaluable Population: all participants who received at least 1 dose of study drug and have provided a Baseline and at least 1 post-dose PK sample
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Groups:
- All Participants: Participants with recurrent, advanced locoregional disease or distant metastatic disease who did not receive any prior chemotherapy received retifanlimab 500 mg, administered by IV infusion over 60 minutes on Day 1 Q4W.
Arm/Group | All Participants
Number analyzed (Participants) | 102
micrograms per milliliter (μg/mL) | 144 (32.6)

8. Secondary Outcome: First-dose Cmin of Retifanlimab
Description: Cmin was defined as the minimum observed plasma concentration over the dose interval.
Time Frame: preinfusion, 10 minutes postinfusion (± 10 minutes), and 4 hours postinfusion (± 10 minutes) on Day 1 of Cycle 1
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | All Participants
Number analyzed (Participants) | 102
μg/mL | 20.5 (7.23)

9. Secondary Outcome: First-dose AUC0-t of Retifanlimab
Description: AUC0-t was defined as the area under the plasma concentration-time curve from time zero to time t.
Time Frame: preinfusion, 10 minutes postinfusion (± 10 minutes), and 4 hours postinfusion (± 10 minutes) on Day 1 of Cycle 1
Population: PK Evaluable Population
Measure: Mean (Standard Deviation); unit: day*mg/L
Arm/Group | All Participants
Number analyzed (Participants) | 102
day*mg/L | 1770 (549)

ADVERSE EVENTS:
Time Frame: Deaths were assessed for up to 60.4 months. Adverse events were assessed for up to 846 days (up to approximately 2.3 years).
Description: Treatment-emergent adverse events (TEAEs), defined as either AEs reported for the first time or worsening of pre-existing events after the first dose of study drug until 90 days after the last dose of study drug, are reported for members of the Safety Evaluable Population (all enrolled participants who received at least 1 dose of study drug). AEs with onset on/after starting a new anticancer therapy were not summarized as TEAEs.
Groups:
- Total: Total
Arm/Group | Chemotherapy: Naïve | Chemotherapy: Refractory | Total
All-Cause Mortality (participants affected / at risk) | 39/101 | 3/6 | 42/107
Serious Adverse Events (participants affected / at risk) | 26/101 | 2/6 | 28/107
Other Adverse Events (participants affected / at risk) | 83/101 | 5/6 | 88/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy: Naïve (N=101) | Chemotherapy: Refractory (N=6) | Total (N=107)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 3 (3) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 4 (4) | 0 (0) | 4 (4)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Concomitant disease progression (General disorders) | 1 (1) | 0 (0) | 1 (1)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (2) | 0 (0) | 1 (2)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Eosinophilic fasciitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (2)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (3) | 0 (0) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy: Naïve (N=101) | Chemotherapy: Refractory (N=6) | Total (N=107)
Alanine aminotransferase increased (Investigations) | 8 (8) | 0 (0) | 8 (8)
Amylase increased (Investigations) | 8 (11) | 0 (0) | 8 (11)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 1 (1) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (23) | 2 (5) | 19 (28)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 1 (1) | 7 (7)
Asthenia (General disorders) | 19 (24) | 2 (3) | 21 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 7 (7)
Blood creatinine increased (Investigations) | 7 (7) | 1 (1) | 8 (8)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 10 (11) | 0 (0) | 10 (11)
Conjunctivitis (Infections and infestations) | 5 (5) | 1 (1) | 6 (6)
Constipation (Gastrointestinal disorders) | 12 (13) | 0 (0) | 12 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 0 (0) | 10 (11)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 19 (33) | 1 (1) | 20 (34)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 0 (0) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 4 (6) | 1 (1) | 5 (7)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Fatigue (General disorders) | 10 (12) | 3 (3) | 13 (15)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 7 (7) | 1 (1) | 8 (8)
Hyperthyroidism (Endocrine disorders) | 6 (6) | 0 (0) | 6 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (6) | 1 (1) | 2 (7)
Hypophysitis (Endocrine disorders) | 1 (1) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 3 (3)
Hypothyroidism (Endocrine disorders) | 8 (8) | 2 (2) | 10 (10)
Insomnia (Psychiatric disorders) | 6 (6) | 0 (0) | 6 (6)
Lipase increased (Investigations) | 9 (11) | 0 (0) | 9 (11)
Low density lipoprotein increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (3) | 7 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (11) | 3 (3) | 13 (14)
Oedema peripheral (General disorders) | 7 (7) | 0 (0) | 7 (7)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 5 (5)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (26) | 1 (1) | 23 (27)
Pyrexia (General disorders) | 11 (14) | 2 (5) | 13 (19)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 0 (0) | 7 (8)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 1 (1) | 5 (5)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (9) | 1 (1) | 6 (10)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT03599713/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/13/NCT03599713/SAP_001.pdf